CLINICAL TRIAL: NCT06741865
Title: Intervention Strategies for Preserving Intellectual Resilience and Engagement
Brief Title: The INSPIRE Study: Intervention Strategies for Preserving Intellectual Resilience and Engagement
Acronym: INSPIRE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Healthy Minds Initiative (Other)
Collaborators: American College of Lifestyle Medicine (Other); Charles Drew University of Medicine and Science (Other); University of California, Los Angeles (Other); Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20211795
Record Dates: First submitted 2024-08-12; First posted 2024-12-19 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Dementia
Keywords: Dementia; Alzheimer
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: The INSPIRE Study is a randomized controlled trial (RCT) with 2,000 participants aged 55 and older. Participants will be randomly assigned to either an intervention group, receiving a personalized, lifestyle-based program with health coaching, or a control group, receiving standard health education materials. Both groups will undergo baseline and follow-up assessments, including cognitive tests and lifestyle evaluations. The study emphasizes community engagement and culturally relevant interventions, aiming to provide insights into the impact of lifestyle changes on cognitive health and to inform public health strategies for dementia prevention in at-risk populations.
Who Masked: Participant, Care Provider
Masking Description: The INSPIRE Study employs a single-blind design, where participants are unaware of their group assignment (intervention or control) to minimize bias in reporting and behavior. However, the investigators and study staff administering the interventions and conducting assessments are not blinded due to the nature of the intervention, which requires direct interaction and coaching. To further reduce potential bias, outcome assessors involved in data analysis will remain blinded to the group assignments until after the primary data analysis is completed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lifestyle Intervention (Experimental): This arm involves an active intervention with health coaching and lifestyle changes.
  Interventions: Behavioral: Lifestyle Intervention
- Standard Health Education (Active Comparator): This arm receives a standard educational approach without the intensive intervention.
  Interventions: Other: Standard Health Education

INTERVENTIONS:
Behavioral: Lifestyle Intervention — This arm involves interventions like health coaching, dietary changes, exercise programs, and other lifestyle modifications.
  Arms: Lifestyle Intervention
Other: Standard Health Education — Participants in the Standard of Care Arm will receive basic educational materials focused on general cognitive and physical health maintenance.
  Arms: Standard Health Education

SUMMARY:
The INSPIRE Study, initiated by the Healthy Minds Initiative, is a community-based research project aimed at demonstrating the impact of lifestyle factors on cognitive health and the prevention of dementia. Conducted in collaboration with the American College of Lifestyle Medicine, Charles Drew University, UCLA, Stanford University and Crenshaw Christian Center, this study focuses on African American communities that are disproportionately affected by lifestyle-dependent diseases. The study involves 2,000 participants aged 55 and older and aims to directly address these disparities by implementing targeted interventions to enhance cognitive function and overall brain health.

DETAILED DESCRIPTION:
The INSPIRE Study, led by the Healthy Minds Initiative, is a groundbreaking community-based research project aimed at exploring the relationship between lifestyle factors and cognitive health, with an emphasis on nutrition and dietary intervention, to prevent dementia and cognitive impairment in African American communities. This study will take place in South Los Angeles, California, a region characterized by significant health disparities, particularly in the prevalence of lifestyle-dependent diseases.

The study, slated to begin in January/February 2025, will involve 2,000 participants aged 55 and older, recruited through community outreach, health education programs, and referrals from local healthcare providers. Participants will undergo a comprehensive initial assessment, including evaluations of medical history, cognitive function, lifestyle habits, and access to health resources.

Participants will be randomized into two groups: an intervention group and a control group. The intervention group will receive personalized guidance from health coaches, participate in an online community forum designed to teach about nutrition and lifestyle risk factor management, and have access to tailored exercise programs, educational materials, and other resources designed to promote cognitive health. The control group will receive standard-of-care educational material and monthly communications aimed at maintaining or improving health. Both groups will undergo baseline assessments and periodic evaluations throughout the study to measure the impact of the interventions on cognitive health.

The study is designed to be culturally relevant and accessible, leveraging community partnerships with organizations such as the American College of Lifestyle Medicine, Charles Drew University, UCLA, Stanford University and Crenshaw Christian Center. These partnerships provide the necessary infrastructure, expertise, and community trust to ensure the study's success.

The INSPIRE Study's primary goal is to demonstrate how targeted lifestyle interventions can reduce the risk of cognitive decline in a population that is particularly vulnerable to such outcomes. By addressing factors such as diet, physical activity, stress management, and social engagement, and management of vascular risk factors, the study aims to create a model for improving brain health that can be replicated in other communities.

The study's findings will not only contribute to the scientific understanding of lifestyle-related cognitive health but also have the potential to inform public health strategies and policy decisions aimed at reducing health disparities. The long-term vision is to establish the Healthy Minds Initiative as a leader in brain health equity, with the INSPIRE Study serving as a blueprint for future interventions.

ELIGIBILITY:
Inclusion Criteria:

* Age: Participants must be 55 years of age or older.
* Ethnicity: Focused on African American individuals, but not exclusive.
* Cognitive Status: Participants must have normal cognitive status, mild cognitive impairment (MCI), or subjective cognitive impairment (SCI).
* Language: Participants must be fluent in English.
* Location: Must reside in the Crenshaw, California area or be able to attend study-related activities in this location.
* Willingness to Participate: Participants must be willing to adhere to the study protocol, including attending assessments, participating in interventions, and completing questionnaires.

Exclusion Criteria:

* Cognitive Decline: Diagnosis of dementia or severe cognitive impairment that would interfere with the ability to participate in the study.
* Physical Limitations: Any physical or medical condition that would preclude participation in the lifestyle interventions (e.g., severe mobility issues).
* Recent Cancer Diagnosis: Diagnosis of cancer within the last three years, excluding stable cases of basal cell or squamous cell carcinoma of the skin, or stable prostate cancer.
* Pregnancy: Current pregnancy or planning to become pregnant during the study period.
* Mental Health: Diagnosis of severe psychiatric disorders such as schizophrenia or bipolar disorder that might interfere with participation.
* Substance Abuse: Current substance abuse or dependency that could impact participation.
* Hearing Impairment: Uncorrected hearing loss that would limit the ability to communicate and participate in the study.
* Non-English Speaking: Inability to participate in English-language oral and written cognitive assessments.
* Participation in Another Study: Currently enrolled in another clinical trial that could interfere with the INSPIRE Study.
* Life expectancy less than 3 years
* Unwillingness to share medical and laboratory information.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-10-13 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Cognitive Function | 6 months, 1 year and 3 years
  Change in global composite score from baseline, as measured by the TABCAT (Tablet-based Cognitive Assessment Tool) composite score, at the designated endpoint (e.g., 6 months, 1 year, and 3 years). This composite score reflects core domains of cognition-including memory, executive function, language, and processing speed-captured through standardized TABCAT assessments.

SECONDARY OUTCOMES:
Adherence to Lifestyle Interventions | Continuous, with key evaluations at 6 months and 12 months.
  Measure adherence to prescribed diet and exercise changes through self-reported questionnaires and logs maintained by health coaches.

OTHER OUTCOMES:
Change in Blood Pressure | 6 months, 1 year and 3 years
  Evaluate changes in blood pressure, as measured by sphygmomanometer at baseline, and then at 6 months, 1 year and 3 years.
Change in Low Density Lipoprotein (LDL) cholesterol levels | 6 months, 1 year and 3 years
  Evaluate changes in Low Density Lipoprotein, as measured by a lipid panel serum test at baseline, and then at 6 months, 1 year and 3 years.
Change in Hemoglobin A1c markers | 6 months, 1 year and 3 years
  Evaluate changes in serum Hemoglobin A1c, a marker of glucose metabolism dysfunction, as measured in the serum, at baseline and then at 6 months, 1 year and 3 years.
Executive functions composite | 6 months, 1 year and 3 years
  Composite score of executive function cognitive test, as measured by TABCAT.
Episodic Memory Composite | 6 months, 1 year and 3 years
  Composite score of episodic memory cognitive test, as measured by TABCAT.

CONTACTS AND LOCATIONS:
Overall Officials: Dean Sherzai, MD, PhD, Principal Investigator — Healthy Minds Initiative
Locations (1):
- Crenshaw Christian Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Livingston G, Huntley J, Liu KY, Costafreda SG, Selbaek G, Alladi S, Ames D, Banerjee S, Burns A, Brayne C, Fox NC, Ferri CP, Gitlin LN, Howard R, Kales HC, Kivimaki M, Larson EB, Nakasujja N, Rockwood K, Samus Q, Shirai K, Singh-Manoux A, Schneider LS, Walsh S, Yao Y, Sommerlad A, Mukadam N. Dementia prevention, intervention, and care: 2024 report of the Lancet standing Commission. Lancet. 2024 Aug 10;404(10452):572-628. doi: 10.1016/S0140-6736(24)01296-0. Epub 2024 Jul 31. No abstract available. PMID 39096926
- [Background] Schippinger WM, Pichler G. [Prevention of dementia]. Z Gerontol Geriatr. 2023 May;56(3):227-234. doi: 10.1007/s00391-023-02175-2. Epub 2023 Apr 25. German. PMID 37097299
- [Background] Willroth EC, Pfund GN, Rule PD, Hill PL, John A, Kyle K, Hassenstab J, James BD. A review of the literature on wellbeing and modifiable dementia risk factors. Ageing Res Rev. 2024 Aug;99:102380. doi: 10.1016/j.arr.2024.102380. Epub 2024 Jun 14. PMID 38880341
- [Background] Dominguez LJ, Veronese N, Vernuccio L, Catanese G, Inzerillo F, Salemi G, Barbagallo M. Nutrition, Physical Activity, and Other Lifestyle Factors in the Prevention of Cognitive Decline and Dementia. Nutrients. 2021 Nov 15;13(11):4080. doi: 10.3390/nu13114080. PMID 34836334
- [Background] Ward DD, Ranson JM, Wallace LMK, Llewellyn DJ, Rockwood K. Frailty, lifestyle, genetics and dementia risk. J Neurol Neurosurg Psychiatry. 2022 Apr;93(4):343-350. doi: 10.1136/jnnp-2021-327396. Epub 2021 Dec 21. PMID 34933996
- [Background] Dhana K, Evans DA, Rajan KB, Bennett DA, Morris MC. Healthy lifestyle and the risk of Alzheimer dementia: Findings from 2 longitudinal studies. Neurology. 2020 Jul 28;95(4):e374-e383. doi: 10.1212/WNL.0000000000009816. Epub 2020 Jun 17. PMID 32554763
- [Background] Low LF, Barcenilla-Wong A, Fitzpatrick M, Swaffer K, Brodaty H, Hancock N, McLoughlin J, Naismith S. Dementia lifestyle coach pilot program. Australas J Ageing. 2023 Sep;42(3):508-516. doi: 10.1111/ajag.13169. Epub 2022 Dec 22. PMID 36546406
- [Background] Aranda MP, Kremer IN, Hinton L, Zissimopoulos J, Whitmer RA, Hummel CH, Trejo L, Fabius C. Impact of dementia: Health disparities, population trends, care interventions, and economic costs. J Am Geriatr Soc. 2021 Jul;69(7):1774-1783. doi: 10.1111/jgs.17345. PMID 34245588
- [Background] Liu C, Murchland AR, VanderWeele TJ, Blacker D. Eliminating racial disparities in dementia risk by equalizing education quality: A sensitivity analysis. Soc Sci Med. 2022 Nov;312:115347. doi: 10.1016/j.socscimed.2022.115347. Epub 2022 Sep 12. PMID 36162365
- [Background] Lennon JC, Aita SL, Bene VAD, Rhoads T, Resch ZJ, Eloi JM, Walker KA. Black and White individuals differ in dementia prevalence, risk factors, and symptomatic presentation. Alzheimers Dement. 2022 Aug;18(8):1461-1471. doi: 10.1002/alz.12509. Epub 2021 Dec 2. PMID 34854531
- [Background] Sherzai D, Sherzai A, Lui K, Pan D, Chiou D, Bazargan M, Shaheen M. The Association Between Diabetes and Dementia Among Elderly Individuals: A Nationwide Inpatient Sample Analysis. J Geriatr Psychiatry Neurol. 2016 May;29(3):120-5. doi: 10.1177/0891988715627016. Epub 2016 Feb 9. PMID 26862150
- [Background] Sherzai D, Sherzai A. Preventing Alzheimer's: Our Most Urgent Health Care Priority. Am J Lifestyle Med. 2019 May 9;13(5):451-461. doi: 10.1177/1559827619843465. eCollection 2019 Sep-Oct. PMID 31523210
- [Background] Morris MC, Tangney CC, Wang Y, Sacks FM, Barnes LL, Bennett DA, Aggarwal NT. MIND diet slows cognitive decline with aging. Alzheimers Dement. 2015 Sep;11(9):1015-22. doi: 10.1016/j.jalz.2015.04.011. Epub 2015 Jun 15. PMID 26086182
- [Background] Barnes LL, Dhana K, Liu X, Carey VJ, Ventrelle J, Johnson K, Hollings CS, Bishop L, Laranjo N, Stubbs BJ, Reilly X, Agarwal P, Zhang S, Grodstein F, Tangney CC, Holland TM, Aggarwal NT, Arfanakis K, Morris MC, Sacks FM. Trial of the MIND Diet for Prevention of Cognitive Decline in Older Persons. N Engl J Med. 2023 Aug 17;389(7):602-611. doi: 10.1056/NEJMoa2302368. Epub 2023 Jul 18. PMID 37466280
- [Background] Morris MC, Tangney CC, Wang Y, Sacks FM, Bennett DA, Aggarwal NT. MIND diet associated with reduced incidence of Alzheimer's disease. Alzheimers Dement. 2015 Sep;11(9):1007-14. doi: 10.1016/j.jalz.2014.11.009. Epub 2015 Feb 11. PMID 25681666
- [Background] McLeod A, Bernabe BP, Xia Y, Sanchez-Flack J, Lamar M, Schiffer L, Hemphill NO, Fantuzzi G, Maki P, Fitzgibbon M, Tussing-Humphreys L. Exploring the Effects of a Mediterranean Diet and Weight Loss on the Gut Microbiome and Cognitive Performance in Older, African American Obese Adults: A Post Hoc Analysis. Nutrients. 2023 Jul 27;15(15):3332. doi: 10.3390/nu15153332. PMID 37571270